CLINICAL TRIAL: NCT01317277
Title: Personalized Text Messages to Improve ART Adherence in HIV+ Methamphetamine Users
Brief Title: Personalized Text Messages to Improve Antiretroviral Treatment (ART) Adherence in HIV+ Methamphetamine Users
Acronym: iTAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, David J. Moore, Ph.D., Associate Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R34DA031058-01A1 (NIH)
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: HIV; AIDS
Keywords: interventions; technology; drug abuse; methamphetamine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personalized Reminder Texting (iTAB) + Psychoeducation (Experimental): Participants in the individualized Texting for Adherence Building (iTAB) arm will receive daily text messaging reminders for antiretroviral medication adherence. These text messages will be targeted to the specific schedule and needs of the individual. Participants will also receive a one-time psychoeducational intervention reviewing the importance of adherence to anti-HIV medications.
  Interventions: Behavioral: individualized Texting for Adherence Building (iTAB)
- Psychoeducation (CTRL) (Active Comparator): Participants will receive a one-time psychoeducational intervention reviewing the importance of adherence to anti-HIV medications. They will also receive daily text messages to evaluate mood and methamphetamine use, but these messages will not remind participants about medication adherence.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: individualized Texting for Adherence Building (iTAB) — Behavioral: Psychoeducation
  Participants will also receive daily text messages to evaluate mood and methamphetamine use, but these messages will not remind participants about medication adherence.
  Behavioral: individualized Texting for Adherence Building (iTAB)
  Intervention is designed to send automated text messages to HIV+ persons who are current methamphetamine (METH+) users. Text messages are personalized, automated, real-time text messages. The iTAB intervention is designed to improve adherence to ART medications among HIV+/METH+ persons above and beyond an active comparator group.
  Arms: Personalized Reminder Texting (iTAB) + Psychoeducation
Behavioral: Psychoeducation — Behavioral: Psychoeducation
  Participants will also receive daily text messages to evaluate mood and methamphetamine use, but these messages will not remind participants about medication adherence.
  Arms: Psychoeducation (CTRL)

SUMMARY:
Methamphetamine (METH) is a debilitating and frequently abused substance that is often comorbid with HIV infection. HIV+ persons with current METH abuse or dependence (HIV+/METH+) have several characteristics, in addition to their substance use, that make them particularly susceptible to nonadherence to antiretroviral treatment (ART) including elevated rates of neurocognitive impairment, co-occurrence of psychiatric disorders, and unstable living situations. The investigators propose an intervention development study designed to address these potential mechanisms of nonadherence with the following Specific Aims: 1) To further develop and refine a personalized, automated, real-time, mobile phone, text messaging intervention (iTAB) designed to improve adherence to ART medications among HIV+/METH+ persons; 2) To evaluate the acceptability and effectiveness of a brief psychoeducation plus text messaging intervention (iTAB) as compared to psychoeducation alone (CTRL) for the improvement of objectively measured medication adherence among HIV+/METH+ persons; and 3) To examine predictors of within-person trajectories of nonadherence using the longitudinal data collected over the study. In order to realize these aims, the investigators will leverage the infrastructure of two unique UCSD resources increasing likelihood of study success, impact, and innovation: 1) the Translational Methamphetamine AIDS Research Center (TMARC), which is a NIDA-funded center that focuses on the combined effects of METH and HIV infection, and 2) the California Institute for Telecommunications and Information Technology (Calit2), which conducts research on state-of-the-art wireless means of health promotion. Initially, the investigators will refine the iTAB intervention to ensure that it is user-centered and tailored to the needs of HIV+/METH+ persons via focus groups and rapid prototyping. Once refined, the proposed iTAB intervention will use text messages that are automated, scalable, personalized, interactive, flexible, and motivating. The investigators will assess the acceptability and effectiveness of iTAB in improving objectively measured adherence (i.e., MEMS caps) over a 6-week period via a pilot RCT with 40 HIV+/METH+ assigned to the iTAB intervention and 20 HIV+/METH+ assigned to a psychoeducational control. Predictors of nonadherence including frequency of METH use, neuropsychological impairment, and mood will be examined to determine whether iTAB is better able to compensate for these factors associated with nonadherence as compared to CTRL. Further refinement to the iTAB intervention will be made in order to pursue a large-scale R01 using our tailored intervention.

ELIGIBILITY:
Inclusion/exclusion criteria are generally lenient in order to ensure that our sample is as representative as possible of the overall HIV+/METH+ population.

Inclusion Criteria:

* Ability to provide informed consent
* 18 years or older at the time of enrollment
* HIV-infected
* DSM-IV diagnosis of methamphetamine abuse or dependence in the past 30 days
* Taking at least one medication to treat HIV illness
* Indication of less than 100% adherence to antiretroviral (ART) medication
* Willingness to use electronic monitoring caps to track ART medication
* Willingness to respond to text messages

Exclusion Criteria:

* Axis I psychiatric diagnosis of psychotic disorder or mood disorder with psychotic features
* Presence of a neurological condition (beyond HIV infection) known to impact cognitive functioning (e.g., Huntington's Disease, Stroke)
* Unwillingness or inability to use electronic medication monitoring technology
* Unwillingness or inability to use daily text messaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Moore, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- Hnrc-Tmarc, San Diego, California, United States

REFERENCES:
- [Result] Moore DJ, Pasipanodya EC, Umlauf A, Rooney AS, Gouaux B, Depp CA, Atkinson JH, Montoya JL. Individualized texting for adherence building (iTAB) for methamphetamine users living with HIV: A pilot randomized clinical trial. Drug Alcohol Depend. 2018 Aug 1;189:154-160. doi: 10.1016/j.drugalcdep.2018.05.013. Epub 2018 Jun 21. PMID 29958127
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Moore DJ, Montoya JL, Blackstone K, Rooney A, Gouaux B, Georges S, Depp CA, Atkinson JH, Tmarc Group T. Preliminary Evidence for Feasibility, Use, and Acceptability of Individualized Texting for Adherence Building for Antiretroviral Adherence and Substance Use Assessment among HIV-Infected Methamphetamine Users. AIDS Res Treat. 2013;2013:585143. doi: 10.1155/2013/585143. Epub 2013 Sep 3. PMID 24078868

RESULTS

PARTICIPANT FLOW:
Groups:
- iTAB + Psychoeducation: individualized Texting for Adherence Building (iTAB): Participants will receive daily text messaging reminders for antiretroviral medication adherence. These text messages will be targeted to the specific schedule and needs of the individual. Participants will also receive daily text messages to assess mood and methamphetamine use.
  Participants will receive a one-time psychoeducational intervention reviewing the importance of adherence to anti-HIV medications.
- Psychoeducation: Participants will receive a one-time psychoeducational intervention reviewing the importance of adherence to anti-HIV medications.
  Participants will also receive daily text messages to evaluate mood and methamphetamine use, but these messages will not remind participants about medication adherence.
Period: Overall Study
Arm/Group | iTAB + Psychoeducation | Psychoeducation
Started | 50 | 25
Completed | 43 | 23
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Lost MEMS | 1 | 1
Not completed — Unable to comply with intervention | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: 371 participants were assessed for eligibility. Of the 75 participants allocated to study group (50 in iTAB, 25 in active control), 68 participants completed follow-up visits (44 in iTAB, 24 in active control group); 1 participant in each study arm was excluded from analyses due to loss of MEMS. 66 participants were included in analyses (43 in iTAB group, 23 in active control group)
Groups:
- Total: Total of all reporting groups
Arm/Group | iTAB + Psychoeducation | Psychoeducation | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 371 participants were assessed for eligibility. Of the 75 participants allocated to study group (50 in iTAB, 25 in active control), 68 participants completed follow-up visits (44 in iTAB, 24 in active control group); 1 participant in each study arm was excluded from analyses due to loss of MEMS. 66 participants were included in analyses (43 in iTAB group, 23 in active control group)
  years
    number analyzed (Participants) | 43 | 23 | 66
    (all) | 45.4 (7.7) | 46.0 (8.9) | 45.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 371 participants were assessed for eligibility, of which 50 (iTAB) and 25 (active control) were allocated; 66 participants completed follow-up (42 iTAB, 24 control); 1 participant was excluded from analyses in each group for losing MEMS. 66 participants were included in analyses (43 in iTAB group, 23 in active control group)
  Participants
    number analyzed (Participants) | 43 | 23 | 66
    Female | 3 | 0 | 3
    Male | 40 | 23 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 371 participants were assessed for eligibility. Of the 75 participants allocated to study group (50 in iTAB, 25 in active control), 68 participants completed follow-up visits (44 in iTAB, 24 in active control group); 1 participant in each study arm was excluded from analyses due to loss of MEMS. 66 participants were included in analyses (43 in iTAB group, 23 in active control group)
  Participants
    Non-Hispanic White: number analyzed (Participants) | 43 | 23 | 66
    Non-Hispanic White | 23 | 7 | 30
    Non-Hispanic Black: number analyzed (Participants) | 43 | 23 | 66
    Non-Hispanic Black | 15 | 7 | 22
    Hispanic: number analyzed (Participants) | 43 | 23 | 66
    Hispanic | 5 | 8 | 13
    Pacific Islander: number analyzed (Participants) | 43 | 23 | 66
    Pacific Islander | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Overall MEMS Adherence to Antiretroviral Medication
Description: Adherence was defined as the percentage of taken doses using Medication Event Monitoring Systems (MEMS); i.e., [(# of bottle openings)/(# of prescribed doses)*100].
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of taken doses
Groups:
- iTAB + Psychoeducation: Participants in the individualized Texting for Adherence Building (iTAB) arm will receive daily text messaging reminders for antiretroviral medication adherence. These text messages will be targeted to the specific schedule and needs of the individual. Participants will also receive a one-time psychoeducational intervention reviewing the importance of adherence to anti-HIV medications.
  individualized Texting for Adherence Building (iTAB): Intervention is designed to send automated text messages to HIV+ persons who are current methamphetamine (METH+) users. Text messages are personalized, automated, real-time text messages. The iTAB intervention is designed to improve adherence to ART medications among HIV+/METH+ persons above and beyond an active comparator group.
- Psychoeducation: Participants will receive a one-time psychoeducational intervention reviewing the importance of adherence to anti-HIV medications. They will also receive daily text messages to evaluate mood and methamphetamine use, but these messages will not remind participants about medication adherence.
  Psychoeducation: Participants will also receive daily text messages to evaluate mood and methamphetamine use, but these messages will not remind participants about medication adherence.
Arm/Group | iTAB + Psychoeducation | Psychoeducation
Number analyzed (Participants) | 43 | 23
percentage of taken doses | 68.0 (0.3) | 70.4 (0.3)
Statistical Analysis 1: Comparison: iTAB + Psychoeducation vs Psychoeducation; Randomization strategy for target 75 participants of 2:1 [iTAB(n=50):CTRL(n=25)], resulting in 80% power to detect effect size of .71 for difference of adherence rates between groups (Wilcoxon-Mann-Whitney critical t=1.99, df=69.6). Final # analyzed: iTAB (n=43) & CTRL (n=23); Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — In between-group analyses, overall MEMS adherence was defined as % of doses taken; Non-parametric methods

2. Primary Outcome: MEMS Adherence to Antiretroviral Medication Based on Dose Timing
Description: Adherence using Medication Event Monitoring Systems (MEMS) based on dose timing; i.e., [(# of bottle openings within a +/- 2-hour time window of the intended dosing time)/(# of prescribed doses)*100].
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of taken doses
Arm/Group | iTAB + Psychoeducation | Psychoeducation
Number analyzed (Participants) | 43 | 23
percentage of taken doses | 43.9 (32.2) | 45.5 (30.5)
Statistical Analysis 1: Comparison: iTAB + Psychoeducation vs Psychoeducation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney) — MEMS adherence based on dose timing was examined for between-group differences; Non-parametric methods

3. Secondary Outcome: Text-reported METH Use
Description: For each participant, we calculated the responsiveness to texts assessing METH use [i.e., (# of texts responded to)/(# of texts received)], and proportion of days a participants endorsed METH use [i.e., (# of days endorsing METH use)/(# of texts responded to)].
Time Frame: Completion of 6-week intervention
Measure: Mean (Inter-Quartile Range); unit: METH use days
Arm/Group | iTAB + Psychoeducation | Psychoeducation
Number analyzed (Participants) | 43 | 23
METH use days | 14.4 [0 to 33.6] | 22.0 [7.3 to 65.6]
Statistical Analysis 1: Comparison: iTAB + Psychoeducation; Text-reported METH use days; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — Z = -1.97; Non-parametric methods; P-Value is calculated

ADVERSE EVENTS:
Arm/Group | iTAB + Psychoeducation | Psychoeducation
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/25
Other Adverse Events (participants affected / at risk) | 1/50 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iTAB + Psychoeducation (N=50) | Psychoeducation (N=25)
Other medical complications (Immune system disorders) | 1 (1) | 0 (0) — Participant developed other medical complications not related to study participation

LIMITATIONS AND CAVEATS:
1) Small sample size; 2) Short time period; 3) MEMS adherence data based on # of cap openings, not directly whether the medication was ingested; 4) No group without psychoeducation component

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No